CLINICAL TRIAL: NCT06419478
Title: Exploring Early Postoperative Core Symptoms in Chinese Patients With Primary Liver Cancer: a Cross-sectional and Longitudinal Network Analysis
Brief Title: Postoperative Symptoms in Chinese Liver Cancer Patients: Network Analysis
Acronym: PSC-LCNA
Status: Terminated | Type: Observational
Why Stopped: The study stopped because recruitment goals were met ahead of schedule.
Sponsor: Mengmeng Yuan (Other)
Collaborators: Anhui Medical University (Other)
Responsible Party: Sponsor-Investigator, Mengmeng Yuan, Research Assistant, Anhui Medical University
Organization: Anhui Medical University (Other)
Other Study IDs: 83242306; 2023AH050604 (Other Grant/Funding Number: the Natural Science Foundation of Anhui Provincial)
Record Dates: First submitted 2024-05-14; First posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Patients With Primary Liver Cancer (PLC) Undergoing Curative Surgical Procedures; Importance of Identifying Core Symptoms for Improving Symptom Management in PLC Patients; Application of Network Analysis as a Crucial Component of Cancer Care
Keywords: Cancer Liver; Hepatectomy; Network analysis; Symptom burden
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- postoperative symptoms: Investigation of postoperative symptoms in eligible patients undergoing liver resection at two time points
  Interventions: Other: postoperative symptoms

INTERVENTIONS:
Other: postoperative symptoms — Observational study, focusing solely on symptom surveys of patients.

SUMMARY:
Patients with primary liver cancer (PLC) experience a range of symptoms in the early postoperative period. Symptoms include cancer-related symptoms and adverse effects of treatment. Exploring the core symptoms and their dynamics in the early post-hepatectomy patients may help provide better symptom management programs. The purpose of this study was to identify the core symptoms in early post-hepatectomy patients and to explore the trajectory of their dynamics. During the period from March 2021 to September 2022, a total of 281 patients diagnosed with PLC and undergoing radical curative surgery were recruited from the hepatobiliary surgery departments of two hospitals in Eastern China, among whom 249 individuals (88.60%) agreed to participate in the study. A comprehensive symptom assessment was administered to the patients 1-2 days after surgery (T1) and 1-2 days before discharge (T2). Network analysis was used to identify core symptoms in early post-hepatectomy patients based on symptom severity.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients were ≥18 years of age; had a diagnosis of primary liver cancer based on pathologic examination; were receiving the first hepatectomy; were conscious, spoke Chinese, and had basic communication skills.

Exclusion Criteria:

* Exclusion criteria include concurrent malignant tumors, mental disorders, or consciousness impairments, as well as participation in other clinical interventions.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with PLC who underwent curative surgical procedures between March 2021 and September 2022 at the Hepatobiliary Surgery Departments of two Eastern Chinese hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 249 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
MD Anderson Symptom Inventory | 1-2 days after surgery (T1) and 1-2 days before discharge (T2).
  The MD Anderson Symptom Inventory (MDASI) is one of the most widely used symptom assessment tools for cancer patients in clinical and research settings and is used to evaluate the severity of symptoms and their impact on daily life. It consists of 13 core symptom items and 6 symptom interference items. The severity of each symptom is rated on an 11-point Likert scale (0 = "not at all" and 10 = "as bad as you can imagine"). The MDASI-C, a Chinese version translated in 2004 by Wang et al., has good reliability, with a Cronbach's alpha of 0.82-0.94.

SECONDARY OUTCOMES:
Symptom Module Specific for Primary Liver Cancer | 1-2 days after surgery (T1) and 1-2 days before discharge (T2).
  The Symptom Module Specific for Primary Liver Cancer (TSM-PLC) can serve as an important supplement to the MDASI, providing instrumental security for the systematic assessment of symptoms in patients PLC. It consists of six symptom items: abdominal distension, diarrhea, loss of weight, jaundice, pruritus, and fever. The six items were rated in the same format as the first part of the MDASI. The TSM-PLC has good reliability (Cronbach's alpha of 0.835 for internal consistency and content validity of 0.91).

CONTACTS AND LOCATIONS:
Overall Officials: shuwen M Li, PhD, Study Chair — Anhui Medical University
Locations (1):
- Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual participant data (Share IPD) to protect participant privacy. However, individuals who support the findings of this study may contact the study's principal investigator directly to request data.

REFERENCES:
- [Background] Zhu Z, Hu Y, Xing W, Guo M, Zhao R, Han S, Wu B. Identifying Symptom Clusters Among People Living With HIV on Antiretroviral Therapy in China: A Network Analysis. J Pain Symptom Manage. 2019 Mar;57(3):617-626. doi: 10.1016/j.jpainsymman.2018.11.011. Epub 2018 Nov 20. PMID 30465875
- [Background] Wang XS, Wang Y, Guo H, Mendoza TR, Hao XS, Cleeland CS. Chinese version of the M. D. Anderson Symptom Inventory: validation and application of symptom measurement in cancer patients. Cancer. 2004 Oct 15;101(8):1890-901. doi: 10.1002/cncr.20448. PMID 15386315
- [Result] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Result] Devarbhavi H, Asrani SK, Arab JP, Nartey YA, Pose E, Kamath PS. Global burden of liver disease: 2023 update. J Hepatol. 2023 Aug;79(2):516-537. doi: 10.1016/j.jhep.2023.03.017. Epub 2023 Mar 27. PMID 36990226
- [Result] Zou H, Li M, Lei Q, Luo Z, Xue Y, Yao D, Lai Y, Ung COL, Hu H. Economic Burden and Quality of Life of Hepatocellular Carcinoma in Greater China: A Systematic Review. Front Public Health. 2022 Apr 21;10:801981. doi: 10.3389/fpubh.2022.801981. eCollection 2022. PMID 35530735
- [Result] Liu D, Song T. Changes in and challenges regarding the surgical treatment of hepatocellular carcinoma in China. Biosci Trends. 2021 Jul 6;15(3):142-147. doi: 10.5582/bst.2021.01083. Epub 2021 Mar 14. PMID 33716267
- [Result] Drott J, Bjornsson B, Sandstrom P, Bertero C. Experiences of Symptoms and Impact on Daily Life and Health in Hepatocellular Carcinoma Patients: A Meta-synthesis of Qualitative Research. Cancer Nurs. 2022 Nov-Dec 01;45(6):430-437. doi: 10.1097/NCC.0000000000001044. Epub 2022 Jan 13. PMID 35025775
- [Result] Ellis J, Brearley SG, Craven O, Molassiotis A. Understanding the symptom experience of patients with gastrointestinal cancers in the first year following diagnosis: findings from a qualitative longitudinal study. J Gastrointest Cancer. 2013 Mar;44(1):60-7. doi: 10.1007/s12029-012-9443-9. PMID 23054580
- [Result] Ryu E, Kim K, Cho MS, Kwon IG, Kim HS, Fu MR. Symptom clusters and quality of life in Korean patients with hepatocellular carcinoma. Cancer Nurs. 2010 Jan-Feb;33(1):3-10. doi: 10.1097/NCC.0b013e3181b4367e. PMID 19926981
- [Result] Patel N, Maher J, Lie X, Gwaltney C, Barzi A, Karwal M, Macarulla T, Sun HC, Trojan J, Meyers O, Workman C, Morgan S, Negro A, Cohen G. Understanding the patient experience in hepatocellular carcinoma: a qualitative patient interview study. Qual Life Res. 2022 Feb;31(2):473-485. doi: 10.1007/s11136-021-02903-4. Epub 2021 Jun 11. PMID 34115280
- [Result] Zhu Z, Sun Y, Kuang Y, Yuan X, Gu H, Zhu J, Xing W. Contemporaneous symptom networks of multidimensional symptom experiences in cancer survivors: A network analysis. Cancer Med. 2023 Jan;12(1):663-673. doi: 10.1002/cam4.4904. Epub 2022 Jun 1. PMID 35651298
- [Result] Cha EJ, Hong S, Park DH, Ryu SH, Ha JH, Jeon HJ. A network analysis of panic symptoms in relation to depression and anxiety sensitivity in patients with panic disorder. J Affect Disord. 2022 Jul 1;308:134-140. doi: 10.1016/j.jad.2022.04.062. Epub 2022 Apr 13. PMID 35429524
- [Result] Zeng L, Huang H, Liu Y, Ruan C, Fan S, Xia Y, Zhou J. The core symptom in multiple myeloma patients undergoing chemotherapy: a network analysis. Support Care Cancer. 2023 Apr 25;31(5):297. doi: 10.1007/s00520-023-07759-7. PMID 37097532
- [Result] Bai W, Cai H, Wu S, Zhang L, Feng KX, Li YC, Liu HZ, Du X, Zeng ZT, Lu CM, Mi WF, Zhang L, Ding YH, Yang JJ, Jackson T, Cheung T, An FR, Xiang YT. Internet addiction and its association with quality of life in patients with major depressive disorder: a network perspective. Transl Psychiatry. 2022 Apr 4;12(1):138. doi: 10.1038/s41398-022-01893-2. PMID 35379778
- [Result] Cleeland CS, Mendoza TR, Wang XS, Chou C, Harle MT, Morrissey M, Engstrom MC. Assessing symptom distress in cancer patients: the M.D. Anderson Symptom Inventory. Cancer. 2000 Oct 1;89(7):1634-46. doi: 10.1002/1097-0142(20001001)89:73.0.co;2-v. PMID 11013380